CLINICAL TRIAL: NCT04277052
Title: Investigation of Masseter and Temporalis Muscles Sections in Individuals With Temporomandibular Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Research Assistant, Physiotherapist, MSc, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2019-112
Record Dates: First submitted 2020-02-16; First posted 2020-02-20 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Joint Disorders; Ultrasonography; Cross sectional
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): Muscle disorders
  Interventions: Device: Determination muscles sections by Ultrasonography
- Group 2 (Experimental): Disc displacements
  Interventions: Device: Determination muscles sections by Ultrasonography
- Group 3 (Experimental): Other common joint disorders
  Interventions: Device: Determination muscles sections by Ultrasonography
- Group 4 (Experimental): Mix type
  Interventions: Device: Determination muscles sections by Ultrasonography
- Group 5 (Experimental): Healthy individuals
  Interventions: Device: Determination muscles sections by Ultrasonography

INTERVENTIONS:
Device: Determination muscles sections by Ultrasonography — Determination muscles sections by Ultrasonography

SUMMARY:
The aim of the study is to examine masseter and temporal muscle sections with Ultrasonography in this individuals depending on the origin of Temporomandibular Disorders.

DETAILED DESCRIPTION:
Multidirectional evaluations are needed to examine the symptoms of Temporomandibular Disorders (TMD). Physical examination, questionnaires towards symptoms, and imaging techniques provide objective data on pathology. The chewing muscles should also be evaluated in this way and the approaches to be followed in subsequent processes should be determined. It is known that muscle sections are changed in TMD, which develops due to muscle disorders. However, regardless of the origin of TMD chewing muscles are affected depending on the condition.

ELIGIBILITY:
Inclusion Criteria:

* Having a temporomandibular disorder,
* Individuals who suited Temporomandibular Disorders/ Research Diagnostic Criteria classification

Exclusion Criteria:

* Pregnant,
* Canser,
* Trauma,
* Neurologic disorder,
* Infection,
* Trigeminal or postherpatic neuralgia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the thickness of the masseter and temporalis muscles sections by Ultrasonography and the changes in the biomechanical properties of the masticatory muscles in individuals with temporomandibular disorders. | Day 1
  US has been described as an accurate and reliable imaging technique to assess the thickness and cross-sectional area of the chewing muscles and to determine changes in the local cross-sectional dimensions of the head and neck muscles in livings. It allows large-scale long-term studies of changes in the thickness of the jaw muscles during the development associated with changes in the biomechanical properties of the masticatory muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Halime ARIKAN, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR